CLINICAL TRIAL: NCT03427320
Title: A Radiopharmacokinetic and Radiodosimetric Phase I/II Imaging Study of 1-alpha-D-(5-[131I]Iodo-5-deoxyarabinofuranosyl)-2-Nitroimidazole (131I-IAZA) in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Imaging of Advanced Tumours Using [131]I-IAZA
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Abandoned.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PK-IAZA-001
Record Dates: First submitted 2017-12-20; First posted 2018-02-09 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2018-02

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: [131]I-IAZA Imaging study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [131]I-IAZA whole body and SPECT imaging (Experimental): Injection of a single dose of 185MBq ( range 150-220MBq) of [131]I-IAZA prior to whole body imaging acquisition at 0-1 hrs,1-3 hrs , 4-8 hrs,19-36 hrs,41-72 hrs and 6-8 days post-injection. SPECT CT of target lesion(s) will be acquired at 19-36 hrs post injection.
  Interventions: Drug: [131]I-IAZA

INTERVENTIONS:
Drug: [131]I-IAZA — Injection of a single dose of 185MBq ( range 150-220MBq) of [131]I-IAZA prior to whole body imaging acquisition at 0-1 hrs,1-3 hrs , 4-8 hrs,19-36 hrs,41-72 hrs and 6-8 days post-injection. SPECT CT of target lesion(s) will be acquired at 19-36 hrs post injection.
  Other Names: 131IAZA

SUMMARY:
Hypoxic cells in tumors have less oxygen than normal cells do, which leads to several changes inside the cells that lead to genetic chages making these cells resistant to treatment. The end result of this is increased tumor growth, spread of the tumor and poor outcome. Early studies have shown that [131]I-IAZA scans can help detect if there are hypoxic cells in the tumor. A [131]I-IAZA scan is a nuclear medicine test used to create pictures of the whole body after [131]I-IAZA is injected into a vein. Further scientific research will help understand how [131]I-IAZA is distributed throughout the body and how it can be used to treat hypoxic tumor cells.

The purpose of this study is to :

1. Demonstrate the safety of [131]I-IAZA
2. To Determine the biodistribution and tumor avidity of [131]I-IAZA in patients with locally advanced or metastatic solid tumors.
3. To determine the optimal imaging time of [131]I-IAZA SPECT.
4. To collect data from imaging and plasma sampling for radiopharmacokinetic analysis of [131]I-IAZA.
5. To determine whole body dosimetry of [131]I-IAZA in selected patients.
6. To evaluate tumor dosimetry of [131]I-IAZA in patients with positive uptake.
7. To determine the radiation dose accrued in hypoxic tumors.

DETAILED DESCRIPTION:
The proposed clinical trial will be a Phase I/II open-label, single site, radiopharmacokinetic and radiodosimetric study in participants with locally advanced or metastatic solid tumors. All participants will be administered oral potassium iodide tablets to block radioactive iodine uptake in the thyroid. After administration of 185 MBq [131]I-IAZA (range: 150 - 220 MBq), all participants will undergo a series of up to six whole body planar scans on a dual headed gamma camera, and blood sampling for radiopharmacokinetic evaluation. A single fecal sample will be collected for up to 5 participants 24 - 72 hours post-injection, if possible, and assessed for total radioactivity. A safety evaluation will be conducted on the first 10 consecutively enrolled participants (safety sub-group), consisting of: Thyroid stimulating hormone (TSH) pre-injection and 6 weeks ±1 week post-injection; vital signs pre-injection and after scans 3 and 4; haematology, and SMA-12 serum biochemistry profile pre-injection and after scans 3 and 4; and an AE assessment at each imaging time point, up to 8 days post-injection. The safety evaluation for the remaining participants will consist of an AE assessment at each imaging time point, up to 8 days post-injection of [131]I-IAZA.

The radiodosimetry of [131]I-IAZA in different tissues will be determined in the first 5 consecutively enrolled participants from the planar images and the measured radioactivity in the fecal samples, if available. SPECT/CT imaging of the tumor(s) will be acquired at 19-36 hours post-injection for all the participants and will be used along with the planar images to determine the radiodosimetry and pattern of dose distribution within the tumor(s). Dosimetry data will be potentially correlated with the participants' health status, or other relevant information, as applicable .

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤ 75 years of age;
* Subjects with locally advanced or metastatic solid tumors with at least one lesion evaluable by CT or magnetic resonance imaging (MRI) of at least 1 cm (smallest diameter), as measured by Response Evaluation Criteria In Solid Tumors (RECIST) within 12 weeks of enrolment;
* Liver function tests (total bilirubin, alanine transaminase (ALT), aspartate transaminase (AST) and alkaline phosphatase) ≤ 5 times the upper limit of normal measured within 2 weeks of enrolment. Serum albumin ≥ 23 g/L within 2 weeks of enrolment;
* Haemoglobin concentration ≥ 90 g/L; white blood cell (WBC) count ≥ 3 x 109/L; platelets ≥ 75 x 109/L measured within 2 weeks of enrolment.
* Serum creatinine ≤ 150 µmol/L, and a calculated (Cockcroft-Gault) or estimated glomerular filtration rate (GFR) of ≥ 50 mL/min measured within 2 weeks of enrolment.
* Eastern Cooperative Oncology Group (ECOG) Performance Scale Score ≤ 2 measured within 2 weeks of enrolment;
* Able and willing to follow instructions and comply with the protocol;
* Ability to provide written informed consent prior to participation in the study.

Exclusion Criteria:

* Systemic therapy for tumors within 2 weeks;
* Prior external beam radiation therapy to the only evaluable lesion
* Existing tracheostomy
* Pregnant or breast feeding
* Previously negative 18F-FAZA uptake of only evaluable lesion(s) within 3 months of enrolment.
* Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.)
* Inability to complete the needed investigational examinations due to other reasons (severe claustrophobia, radiation phobia, etc.)
* Any additional medical condition, serious inter-current illness or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study performance or interpretation .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in vital signs after [131]I-IAZA injection (first 10 patients) | Up to 36 hours post-injection
  Vital signs are measured before injection of [131]I-IAZA and after the third and fourth scans
Change in hematology/SMA-12 serum biochemistry after [131]I-IAZA injection (first 10 patients) | Up to 36 hours post-injection
  Hematology and SMA-12 serum biochemistry will be performed before injection of [131]I-IAZA and after the fourth scan.
Change in TSH level after [131]I-IAZA injection | Before [131]I-IAZA injection and 6 weeks ± 1 week after [131]I-IAZA injection
  TSH blood test will be performed before injection of [131]I-IAZA and 5-7 weeks after [131]I-IAZA injection.
Number of participants with adverse events. | Up to 8 days after [131]I-IAZA injection
  All participants will be evaluated for AE occurrence once [131]I-IAZA has been injected and for the following 8 days during which [131]I-IAZA scans will be acquired

SECONDARY OUTCOMES:
Biodistribution and tumor hypoxia avidity of [131]I-IAZA | Up to 8 days
  Analysis of [131]I-IAZA whole body scans and SPECT-CT for biodistribution of [131]I-IAZA
Radioactivity of blood samples withdrawn at each imaging time point. | Up to 8 days
  Radioactivity will be measured in blood samples collected at each imaging time point.
Estimating the whole body dosimetry of [131]IAZA in selected participants | Up to 8 days
  The radiodosimetry of [131]I-IAZA will be determined by outlining organs of significant uptake on the planar images and determining the dose to each normal organ.
Dose of [131]I-IAZA taken up by the tumor (in mSv/MBq) at each imaging time point in patients with positive uptake. | Up to 8 days
  The tumor activity values will be determined from [131]I-IAZA scans and combined into time-activity curves.
Dose (in mSv/MBq of [131]I-IAZA) to bone marrow | Up to 8 days
  The bone marrow absorbed dose will be calculated using the blood activity and dosimetry data from the [131]I-IAZA whole body scans.
Time to maximum [131]I-IAZA uptake | Up to 8 days
  The activity values of different organs will be determined form [131]I-IAZA scans and combined into time-activity curves.
Clearance characteristics of [131]IAZA | Up to 8 days
  [131]I-IAZA scans will be analyzed for the rate and organs involved in clearance of [131]I-IAZA from the body.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander JB McEwan, MB,FRCPC, Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No